CLINICAL TRIAL: NCT05639777
Title: The Effect of Intranasal Dexmedetomidine Premedication in Children Undergoing Adenotonsillectomy Suffering From Recent Mild Upper Respiratory Tract Infection
Brief Title: Intranasal Dexmedetomidine in Children Undergoing Adenotonsillectomy Suffering From Mild Upper Respiratory Tract Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Eman Ahmed Azzam, Resident of Anesthesia, Surgical Intensive Care and Pain Mrdicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 35355/3/22
Record Dates: First submitted 2022-11-26; First posted 2022-12-06 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Dexmedetomidine; Adenotonsillectomy; Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Dexmedetomidine; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intranasal (Experimental): That will receive intranasal dexmedetomidine (1.5mcg/kg)
  Interventions: Drug: Dexmedetomidine group
- control group (Placebo Comparator): That will receive the same volume of 2 ml of intranasal normal saline
  Interventions: Other: control group

INTERVENTIONS:
Drug: Dexmedetomidine group — That will receive intranasal dexmedetomidine (1.5mcg/kg)
  Other Names: Precedex
  Arms: Intranasal
Other: control group — That will receive the same volume of 2 ml of intranasal normal saline
  Arms: control group

SUMMARY:
The purpose of this study is to detect the efficacy of intranasal dexmedetomidine as a premedication to general anesthesia in pediatric patients with respiratory comorbidities undergoing adenotonsillectomy.

DETAILED DESCRIPTION:
Respiratory comorbidities are associated with an increased incidence of peri-operative respiratory adverse effects (PRAE).

Upper and lower respiratory infections, as well as asthma, are common in children who are scheduled for adenotonsillectomy. When compared to healthy children, children with respiratory ailments have a three-fold increase in PRAEs.

ELIGIBILITY:
Inclusion Criteria:

1. Children with recent mild URI or asthma.
2. aged from 3 to 10 years
3. ASA Physical Status II,
4. undergoing adenotonsillectomy

Exclusion Criteria:

1. Parental refusal of participation
2. Evidence of moderate to severe upper respiratory tract infection at time of presentation on the day of surgery
3. Lower respiratory tract infection
4. Congenital heart diseases
5. Known hypersensitivity to specific anesthetic agent
6. Liver or renal disease

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2022-12-06 (Actual); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
The incidence of peri-operative respiratory adverse effects (PRAE). | From induction to emergence from general anesthesia.
  All PRAE and the time of occurrence (induction, maintenance or emergence) will be recorded.

SECONDARY OUTCOMES:
Sedating effects of this drug. | 15 and 30 min after sedation
  The sedating effects will be measure using Ramsay sedation scale from 1 to 6 as 1 meaning anxious and agitated, restless, or both. and 6 meaning Unresponsive.
Ease of parental separation. | 15 and 30 min after sedation
  Evaluated using a four-point scale. from 1 to 4 as 1 meaning excellent and 4 for poor
Face mask acceptance. | 15 and 30 min after sedation
  Evaluated using a four-point scale. from 1 to 4 as 1 meaning excellent and 4 for poor
Hemodynamic stability | 15 and 30 min after sedation
  hypertension, tachycardia, bradycardia

CONTACTS AND LOCATIONS:
Overall Officials: Ayman A Yousef, Professor, Principal Investigator — Anesthiology' Surgical Intensive care and Pain Medicine; Gehan M Eid, Professor, Principal Investigator — Assistant Professor Anesthiology' Surgical Intensive care and Pain Medicine; Wail E Messbah, Lecturer, Principal Investigator — Anesthiology' Surgical Intensive care and Pain Medicine
Locations (1):
- Eman Ahmed Azzam, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be upon reasonable request from the principle investigator
Supporting Information: Study Protocol, SAP
Time Frame: For one year after completion of the study